CLINICAL TRIAL: NCT02067598
Title: Effects of Scapular Exercise on Patients With Scapulocostal Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mae Fah Luang University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Vitsarut Buttagat, Mae Fah Luang University, Mae Fah Luang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 55218152-3
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Scapular Pain
Keywords: Scapular exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Scapular exercise (Experimental): The participants will receive thirty minutes session of scapular exercise for 12 sessions
  Interventions: Other: scapular exercise
- Control (No Intervention)

INTERVENTIONS:
Other: scapular exercise
  Other Names: The participants will receive thirty minutes session of scapular exercise for 12 sessions
  Arms: Scapular exercise

SUMMARY:
The purpose of this study is to determine the effect of scapular exercise on pain related parameters including pain intensity, 24 hours pain intensity, pressure pain threshold, anxiety and muscle tension in patients with scapulocostal syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age between 18 - 50 years old
3. The participants have experienced spontaneous scapular pain for longer than 12 weeks (chronic) and that at least one trigger point will be present in the scapular region (serratus posterior superior, rhomboid groups, levator scapulae and trapezius muscles). Trigger points will be diagnosed as the presence of focal tenderness in a taut band and with pain recognition (Chatchawan et al., 2005; Tough et al., 2007).
4. The participants will be able to follow instructions.
5. Good communication and cooperation.

Exclusion Criteria:

1. A history of the following diseases or disorders:

* Rotator cuff disease
* Cervical radiculopathy
* Degenerative shoulder joint disease
* Adhesive capsulitis of shoulder

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold as a measure by algometry | 6 Weeks

SECONDARY OUTCOMES:
Pain scores on visual analog scale | 6 weeks
Muscle tension on visual analog scale | 6 weeks
Anxiety on State Anxiety Inventory | 6 weeks
24 hours pain intensity on Visual analog scale | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- School of Health Science, Mae Fah Luang University, Mueang, Changwat Chiang Rai, Thailand